CLINICAL TRIAL: NCT01428635
Title: Eltrombopag for the Management of Thrombocytopenia Associated With Tyrosine Kinase Therapy in Patients With Chronic Myeloid Leukemia (CML) and Myelofibrosis (MF)
Brief Title: Eltrombopag Olamine in Treating Thrombocytopenia in Patients With Chronic Myeloid Leukemia or Myelofibrosis Receiving Tyrosine Kinase Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0319; NCI-2011-03336 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0319 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Primary Myelofibrosis; Thrombocytopenia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (eltrombopag olamine) (Experimental): Patients receive eltrombopag olamine PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eltrombopag Olamine

INTERVENTIONS:
Drug: Eltrombopag Olamine — Given PO
  Other Names: Promacta; SB-497115-GR

SUMMARY:
This phase II/III trial studies how well eltrombopag olamine works in treating thrombocytopenia in patients with chronic myeloid leukemia or myelofibrosis receiving tyrosine kinase inhibitor therapy. Eltrombopag olamine may cause the body to make platelets after receiving treatment for chronic myeloid leukemia or myelofibrosis.

DETAILED DESCRIPTION:
The goal of this clinical research study is learn if eltrombopag can help control or prevent low platelet counts in patients receiving treatment for CML or myelofibrosis. This is an investigational study. Eltrombopag is FDA approved and commercially available for the treatment of patients with low platelet counts. The use of eltrombopag for the treatment of low platelet counts in patients with CML and myelofibrosis is investigational. Eltrombopag will be provided at no cost to you during the study.

If you are found to be eligible to take part in this study, you will receive eltrombopag by mouth 1 time a day. Your dose may be increased every 2 weeks depending on your platelet count response. You should take eltrombopag on an empty stomach. You should not eat for 2 hours before taking eltrombopag. You should wait at least 4 hours between taking eltrombopag and taking other drugs (like antacids), dairy products, juices with calcium added, or supplements containing iron, calcium, aluminum, magnesium, selenium, or zinc.

Up to 39 patients will take part in this study. All will be enrolled at MD Anderson. As of June 6, 2017, the study is closed to new participants.

ELIGIBILITY:
Inclusion Criteria:

* CML patients in chronic phase receiving treatment with any Food and Drug Administration (FDA) approved TKI; or CML patients in accelerated or blastic phase who are considered to be in this phase because of thrombocytopenia or because of clonal evolution and with no other criteria for accelerated/blastic phase or patients with myelofibrosis receiving treatment with FDA approved TKI and with peripheral blood and/or bone marrow blasts =< 10%
* Grade >= 3 thrombocytopenia (platelets < 50 x 10^9/L) after the first 3 months of therapy with the TKI for patients with CML and platelets < 100 x 10^9/L for patients with MF after the first 3 months of therapy; thrombocytopenia must be either recurrent (i.e., second or greater episode of thrombocytopenia) or having required dose reductions of the TKI
* Subject is anticipated to have therapy with TKI continued for >= 3 months
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except for Gilbert's syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN
* Creatinine =< 2 x ULN

Exclusion Criteria:

* CML patients in accelerated or blastic phase except for those who are considered to be in this phase because of thrombocytopenia or because of clonal evolution and with no other criteria for accelerated/blastic phase; or myelofibrosis patients who have transformed to acute leukemia or have >= 10% blasts in peripheral blood and/or in bone marrow
* Thrombocytopenia that is considered to be unrelated to treatment with TKI or accelerated phase as defined above
* Stem cell transplantation within preceding 60 days prior to registration
* Patients with documented active hepatitis B or C infection
* Patients with known bone marrow reticulin fibrosis (>= grade 2) (only applicable to patients with CML)
* Patients with palpable splenomegaly >= 16 cm below coastal margin (only applicable to patients with CML)
* Female subjects who are pregnant or breastfeeding
* Women of childbearing potential are required to have a beta human chorionic gonadotropin (BHCG) serum or urine pregnancy test performed within 7 days prior to first study drug dose; a female of childbearing potential is a sexually mature woman who:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation
* Patients with known risk factors for thromboembolism (e.g. Factor V Leiden mutation, antithrombin III (ATIII) deficiency, Protein C and S deficiency, antiphospholipid syndrome, portal hypertension, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2012 to January 2022
Groups:
- Supportive Care (Eltrombopag Olamine) CML Participants; Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants: Patients receive eltrombopag olamine PO QD in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
Period: Overall Study
Arm/Group | Supportive Care (Eltrombopag Olamine) CML Participants | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants
Started | 15 | 6
Completed | 15 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Care (Eltrombopag Olamine) CML Participants | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 0 | 13
  >=65 years | 2 | 6 | 8
Age, Continuous [Median (Full Range); unit: years] | 46 [29 to 97] | 73 [67 to 82] | 57 [29 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 6 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Platelet Response
Description: The primary endpoint is complete (platelet) response (yes/no). A complete (platelet) response will be defined as a sustained (3 months) platelet count of > 50 x 109/L for patients with CML and > 100 x 109/L for patients with MF and at least a 20% increase in platelet count from baseline.
Time Frame: Up to 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine) CML Participants | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants
Number analyzed (Participants) | 15 | 6
Participants | 12 | 0

2. Secondary Outcome: Number of Participants With a Response to TKI Therapy After Eltrombopag
Description: (CML) : Complete Hematologic Remission : Normalization for 4 weeks of the bone marrow (< 5% blasts) and peripheral blood with WBC within normal institutional limits with no blasts, promyelocytes or myelocytes, and basophils <5%,. Complete cytogenetic response: Ph positive 0%. Partial cytogenetic response: Ph positive 1-35%. Minor cytogenetic response: Ph positive 36-90%. No cytogenetic response: Ph positive 100%. Myelofibrosis : Complete Remission: absence of transfusion or growth factor support: complete resolution of disease-related symptoms/signs including palpable hepatosplenomegaly, hemoglobin > 11 g/dL, platelet count ≥100 x 10^9/L, absolute neutrophil count ≥ 1.0 x 10^9/L. Normal leukocyte differential with disappearance of nucleated red blood cells and immature myeloid cells in peripheral smear, in the absence of splenectomy. Bone marrow histological remission:presence of age-adjusted normocellularity, < 5% myeloblast , osteomyelofibrosis grade </= 1.
Time Frame: Up to 9 years
Population: Zero participants were analyzed in Myelofibrosis Participants as this outcome measure only analyzes those participants who had a platelet response . Zero participants in the Myelofibrosis group had a platelet response, therefore zero participants in this outcome were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine) CML Participants | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants
Number analyzed (Participants) | 12 | 0
Participants | 9 | 0

ADVERSE EVENTS:
Time Frame: Up to 10 years
Arm/Group | Supportive Care (Eltrombopag Olamine) CML Participants | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/6
Serious Adverse Events (participants affected / at risk) | 10/15 | 4/6
Other Adverse Events (participants affected / at risk) | 13/15 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Eltrombopag Olamine) CML Participants (N=15) | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants (N=6)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2)
Flu Like Symptoms (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (3) | 2 (3)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Eltrombopag Olamine) CML Participants (N=15) | Supportive Care (Eltrombopag Olamine) Myelofibrosis Participants (N=6)
Abdominal pain (General disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (9) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema (General disorders) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Eye Disorders (Eye disorders) | 2 (2) | 0 (0)
Eye Infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Flu Like Symptoms (General disorders) | 1 (1) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Thrombosis (Investigations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (2) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 0 (0)
Pain Extremity (General disorders) | 2 (2) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 3 (3) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT01428635/Prot_SAP_000.pdf